CLINICAL TRIAL: NCT00459082
Title: A Pharmacokinetic Study of Dexmedetomine in Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PPRU 10760
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2007-04

CONDITIONS: Cardiac Surgical Procedures
Keywords: Dexmedetomine; Post-operative cardiac surgery

INTERVENTIONS:
Drug: Dexmedetomine

SUMMARY:
Blind randomized trial of a single bolus dose of dexmedetomine followed by a continuous infusion (CIVI) for up to 24 hours in infants who immediately post-operative from cardiac surgery and require tracheal intubation with mechanical ventilation in the post-operative period. Three bolus and infusion dose will be administered to a total of 36 patients.

DETAILED DESCRIPTION:
This clinical trial of three dose rates of dexmedetomine will determine the pharmacokinetics of the drug in infants who remain tracheally intubated postoperatively. An exploratory pharmacodynamic study of a non-invasive device measuring sedation will be performed. Although the pharmacokinetics of dexmedetomine have been described for pediatric patients, the drug disposition in infants has not been well described. A range of doses has been studied, yet there are no reports describing the optimal dose for post-operative pediatric patients. This study will provide data that may allow for improved dosing recommendations in this critically ill population of children.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 1 month, less than or equal to 24 months
* Post-operative from cardiac surgery with tracheal intubation/mechanical ventilation in the immediate post-operative period
* Planned tracheal extubation within 24 hours post-operative period
* Renal function-serum creatine = 1.5 times the ULN for age
* Total bilirubin less than or equal to 1.5 X upper limit of normal (ULN) for age
* SGPT (ALT) ,less than+ 3x upper limit of normal (ULN) for age
* Signed written informed consent

Exclusion Criteria:

* Patients who have received another investigational drug within the past 30 days
* Receiving intermittent or continuous muscle relaxation during study period
* Patients who have a positive blood culture without a subsequent negative culture or other evidence of ongoing serious infection.
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.
* Post-Operative hypotension
* Heart block
* Weight < 5 kg
* Patients who, in the opinion of the investigator, are not appropriate candidates for an investigational drug study.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36
Dates: Start 2004-05; Study Completion 2006-11

PRIMARY OUTCOMES:
Pharmacodynamics: vital signs, cardiac rhythm, oxygen saturation, laboratory evaluations and adverse events will be monitored to determine the safety of dexmedetomine.
Pharmacokinetics: will measure plasma concentrations for dose escalations of dexmedetomine to determine the maximum tolerated dose (MTD).

SECONDARY OUTCOMES:
Pharmacodynamics: The Bispectral Index Scale(BIS) and the University of Michigan sedation scale will be used to measure the level of sedation and dexmedetomine plasma drug concentrations.
Pharmacogenetics: will examine the relationship between genotype, drug exposure and drug response in infants postoperative form cardiac surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States